CLINICAL TRIAL: NCT06830525
Title: Development of a Personalized Growth Hormone Treatment Profile (PGTP) Report for Pediatric Endocrinology
Acronym: PGTP
Status: Completed | Type: Observational
Sponsor: Luis Fernandez Luque (Industry)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor-Investigator, Luis Fernandez Luque, Chief Scientific Officer, Adhera Health, Inc.
Organization: Adhera Health, Inc. (Industry)
Other Study IDs: PGTP
Record Dates: First submitted 2025-01-23; First posted 2025-02-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Growth Hormone Deficiency (GHD)
Keywords: Growth Hormone Disorder; Digital health; pediatric endocrinology; Personalized Growth Hormone Treatment Profile
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — 2-amino-3-cyano-6-methyl-5-(3,4-dimethoxyphenyl)pyridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families with children undergoing growth hormone treatment: The study targets families of children with growth hormone deficiency (GHD) under growth hormone treatment, using a connected injector device that quantifies treatment adherence. We will recruit 40 families, divided into two groups: one group with adherence rates of <85%, and the other group with adherence rates of >85%.
  Interventions: Combination Product: ACDP® and growth hormone treatment

INTERVENTIONS:
Combination Product: ACDP® and growth hormone treatment — A cohort of 40 families of children undergoing growth hormone treatment using a connected injector devices that quantifies treatment adherence will be recruited via the ACDP®, to capture additional data that combine Patient Reported Outcomes and Adherence Data.

SUMMARY:
The goal of this observational study is to learn how to make growth hormone treatment more personalized for children. The main questions it aims to answer are:

* How can information about treatment adherence and patient experiences help improve care?
* What insights can help doctors create treatment plans that are more tailored to each child?

The study will include 40 families of children who are using a connected injector device for their growth hormone treatment. These devices track how often the treatment is taken, and families will also share their experiences through surveys. The information will be used to develop a new tool, similar to tools used in diabetes care, to help doctors create better, personalized treatment plans for children with growth hormone needs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (up to 18 years old) diagnosed with growth hormone deficiency or disorders requiring growth hormone treatment.
* Patients are currently undergoing growth hormone therapy. Includes both naive patients (those newly starting weekly treatment) and those already on treatment.
* Families willing to use connected injector devices and participate in mobile-based psychometrics for the study duration.
* Families are able and willing to regularly provide patient-reported outcomes (PROs) and adherence data through the Adhera®️ Caring Digital Program.
* Participants willing to sign the informed consent form, confirming their understanding of the essential aspects of the study, including the potential risks, benefits and rights as participants.

Exclusion Criteria:

* Families/patients already enrolled in other study protocols, including the use of connected injector devices and participation in mobile-based psychometrics.
* Patients with other significant medical conditions that could interfere with growth hormone treatment or the study's data collection processes.
* Inability to understand or communicate in the language used for data collection and study participation, unless appropriate translation services are available and can be consistently utilized.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample of the study (children and their caregivers) will be recruited from the Pediatric Endocrinology unit at the Miguel Servet Children's University Hospital. This public hospital provides pediatric health attention to the regional area of Zaragoza (Spain), which covers a total of 367.110 inhabitants.
  Families of children undergoing growth hormone therapy and are willing to join a combined intervention.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Develop a Personalized Growth Hormone Treatment Profile (PGTP) | From enrollment to the end of the study at Month 12
  To develop a Personalized Growth Hormone Treatment Profile (PGTP) standard - analogous to the Ambulatory Glucose Profile (AGP) for diabetes care-, integrating diverse data sources to support personalized treatment strategies in pediatric endocrinology.

SECONDARY OUTCOMES:
Adherence to Treatment Using Connected Injector Devices | From enrollment to the end of the study at Month 12
  Automated tracking of injection times and adherence. Adherence will be quantified through connected injector device data, capturing timestamps of each injection and calculating adherence rates.
Physiological Monitoring via Wearable Devices - Sleep Quality | From enrollment to the end of the study at Month 12
  Unit of Measure:
  - Total sleep duration (hours per night). Description: Sleep parameters will be tracked using wearable devices.
Physiological Monitoring via Wearable Devices - Heart Rate | From enrollment to the end of the study at Month 12
  Unit of Measure: Average daily heart rate (beats per minute, bpm). Description: Daily average heart rate recorded through wearable devices.
Physiological Monitoring via Wearable Devices - Physical Activity Metrics | From enrollment to the end of the study at Month 12
  Unit of Measure:
  * Total calories burned per day (kilocalories, kcal).
  * Total steps per day (steps).
  * Total activity time per day (minutes).
  Description: Data will be collected from wearable devices to assess daily physical activity.
Physiological Monitoring via Wearable Devices - Blood Oxygen Levels | From enrollment to the end of the study at Month 12
  Unit of Measure: Daily oxygen saturation percentage (%). Description: Measured through wearable device sensors.
Evaluating Usability of Connected Devices | From enrollment to the end of the study at Month 12
  Outcome Measure: System Usability Scale (SUS) score. Unit of Measure: SUS score (0-100, higher scores indicate better usability). Description: The System Usability Scale (Bangor et al., 2008) is a 10-item scale based on a 5-point Likert scale assessing perceived usability.
Mobile Application Engagement | From enrollment to the end of the study at Month 12
  Outcome Measure: User engagement with the mobile application. Unit of Measure: Frequency of interactions (e.g., number of logins per day/week).
  Description: Engagement will be assessed using mobile user logs, including user profiling metrics based on Hors-Fraile et al. (2018).
Distress Assessment 2 | From enrollment to the end of the study at Month 12
  Distress Thermometer Unit of Measure: Score on a 0-10 scale (higher scores indicate higher distress).
  Description: The Distress Thermometer is a single-item, self-report tool measuring psychological distress on a 0-10 scale.
Distress Assessment 2 | From enrollment to the end of the study at Month 12
  Depression, Anxiety, and Stress Scale - 21 Items (DASS-21) Unit of Measure: Score range 0-63 (higher scores indicate greater distress). Description: The DASS-21 is a 21-item scale measuring general affective distress, including depression, anxiety, and stress, over the past week.
Self-Efficacy Assessment | From enrollment to the end of the study at Month 12
  General Self-Efficacy Scale (GSE) Unit of Measure: Score range 10-40 (higher scores indicate greater self-efficacy).
  Description: The GSE scale measures an individual's belief in their ability to cope with adversity.
Mood Assessment | From enrollment to the end of the study at Month 12
  Positive and Negative Affect Schedule (PANAS)
  Unit of Measure:
  * Positive Affect (PA) score range: 10-50 (higher scores indicate greater positive affect).
  * Negative Affect (NA) score range: 10-50 (higher scores indicate greater negative affect).
  Description: PANAS is a self-report questionnaire measuring two dimensions of mood: positive and negative affect.
Mental Health and Well-Being Assessment | From enrollment to the end of the study at Month 12
  Mental Health Continuum-Short Form (MHC-SF) Unit of Measure: Score range 0-70 (higher scores indicate better mental health).
  Description: The MHC-SF is a 14-item scale assessing emotional, social, and psychological well-being as indicators of positive mental health.
Health-Related Quality of Life (HRQoL) | From enrollment to the end of the study at Month 12
  KIDSCREEN-10 Unit of Measure: Score range 10-50 (higher scores indicate better health-related quality of life).
  Description: The KIDSCREEN-10 is a health-related quality of life measure for children and adolescents, assessing physical, psychological, and social well-being, autonomy, school environment, and peer and family support.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No